CLINICAL TRIAL: NCT01179984
Title: Bard® LifeStent® Vascular Stent Delivery System Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-09-006
Record Dates: First submitted 2010-05-21; First posted 2010-08-11 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTA and study stent (Experimental): Bard® LifeStent® Vascular Stent System
  Interventions: Device: Bard® LifeStent® Vascular Stent System

INTERVENTIONS:
Device: Bard® LifeStent® Vascular Stent System — Stent Implantation

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of a new delivery system for the Bard® LifeStent® Vascular Stent System.

DETAILED DESCRIPTION:
Single-arm, non-randomized, prospective, multi-center study using the Bard® LifeStent® Vascular Stent Delivery System in subjects with lifestyle-limiting claudication or ischemic rest pain that are candidates for percutaneous transluminal angioplasty (PTA) and stenting with lesion(s) in the infra-inguinal segment (superficial femoral artery (SFA) and/or proximal popliteal artery). Subjects will be treated with PTA followed by implantation of the Bard® LifeStent® Vascular Stent.

Clinical follow-up for all subjects will be performed prior to hospital discharge, 30-days, and 12-, 24-, and 36-months post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal representative has been informed of the nature of the evaluation, agrees to its provisions, and has signed the informed consent form (ICF).
2. Subject agrees to comply with the protocol-mandated follow-up procedures and visits.
3. The subject is ≥ 21 years old.
4. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within seven days prior to index procedure. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test.
5. The subject has lifestyle-limiting claudication or ischemic rest pain defined as: Rutherford Category1 2-4 (moderate claudication to ischemic rest pain).
6. The target lesion(s) has angiographic evidence of stenosis or restenosis ≥50% or occlusion (by visual estimate) and is amenable to PTA and stenting.
7. The total treated segment(s) must be ≤ 240 mm.
8. The target vessel reference diameter is ≥4.0 mm and ≤6.5 mm (by visual estimate) and therefore appropriate for treatment with available stent diameters of 6.0 mm and 7.0 mm.
9. There is angiographic evidence of at least one vessel runoff to the foot (at the level of the malleolus).

Exclusion Criteria:

1. The subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with the study follow-up procedure and visits.
2. The subject has claudication or critical limb ischemia described as Rutherford Category1 1 (mild claudication), 5 (minor tissue loss) or 6 (major tissue loss).
3. The subject has a known contraindication (including allergic reaction) or sensitivity to antiplatelet/anticoagulant medications, nickel, titanium or tantalum.
4. The subject has a known sensitivity to contrast media that is not amenable to pretreatment with steroids or/and antihistamines.
5. The subject has a history of bleeding diatheses or coagulopathy.
6. The subject has concomitant renal failure with a creatinine of >2.5 mg/dL.
7. The subject has concomitant hepatic insufficiency, thrombophlebitis, uremia, systemic lupus erythematosus (SLE), or deep vein thrombosis (DVT) at the time of the study procedure.
8. The subject is receiving dialysis or immunosuppressive therapy.
9. The subject is participating in an investigational drug or another investigational device study.
10. The subject has another medical condition, which, in the opinion of the investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than two years.
11. The subject has extensive peripheral vascular disease, which, in the opinion of the investigator, precludes safe insertion of an introducer sheath.
12. The target lesion(s) is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion(s).
13. The subject has angiographic evidence of poor inflow, which would be deemed inadequate to support a vascular bypass graft.
14. The subject is diagnosed with septicemia at the time of the study procedure.
15. Patients with a stent previously implanted into the target vessel.
16. Bilateral disease in the native SFA and/or proximal popliteal artery where both limbs meet the inclusion/exclusion criteria and it is planned to treat both limbs within 30 days. Note: One limb may be enrolled in the study, but only if the second limb is planned to be treated after the 30-day follow-up visit has taken place. The limb that may be enrolled has to be the limb with the more severe lesion and the reasons for treating this specific limb will need to be stated in the CRF.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Herzzentrum Bad Krozingen, Germany
Locations (8):
- Univ. Prof. Dr. Johannes Lammer, Vienna, Austria
- Germany (7):
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Dr. Henrik Schroeder, Berlin
  - Dr. Hans Krankenberg, Hamburg
  - Dr. Rainer Schmiedel, Kaiserslautern
  - Prof. Dr. med. Dietrich Pfeiffer, Leipzig
  - Prof. Dr. Holger Reinecke, Münster
  - Prof. Dr. Gunnar Tepe, Rosenheim

RESULTS

PARTICIPANT FLOW:
Groups:
- PTA and Study Stent: The study population is comprised of subjects who present with lifestyle-limiting claudication or ischemic rest pain that are candidates for PTA and stenting.
Period: Overall Study
Arm/Group | PTA and Study Stent
Started | 76
Completed | 58
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is comprised of subjects who present with lifestyle-limiting claudication or ischemic rest pain that are candidates for PTA and stenting.
Groups:
- Single-Arm: The study population is comprised of subjects who present with lifestyle-limiting claudication or ischemic rest pain that are candidates for PTA and stenting.
Arm/Group | Single-Arm
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 76
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 76

OUTCOME MEASURES:

1. Primary Outcome: Acute Effectiveness: Percentage of Stents With Successful Delivery
Description: Effectiveness:
  Acute effectiveness defined as the successful delivery of the stent with the post-deployment stent length being within 10% of the pre-deployment length.
Time Frame: At implantation (Day 0)
Measure: Mean (95% Confidence Interval); unit: percentage of stents
Units Other Than Participants: Stents
Arm/Group | PTA and Study Stent
Number analyzed (Participants) | 76
Number analyzed (Stents) | 64
percentage of stents | 100 [90 to 100]

2. Primary Outcome: (Safety) Freedom From Occurrence of Death, Amputation and TVR/TLR at 30-days Post-index Procedure.
Description: Safety:
  Freedom from occurrence of death, amputation and TVR/TLR at 30-days post-index procedure.
Time Frame: 30 day follow-up
Population: Freedom from occurrence of death, amputation and TVR/TLR at 30-days post-index procedure.
Measure: Number; unit: percentage of freedom from events
Arm/Group | Single-Arm
Number analyzed (Participants) | 76
percentage of freedom from events | 75

3. Secondary Outcome: Primary Target Lesion Patency
Description: Percentage of participants with Primary Target Lesion Patency (TLP) at 12 months post-index procedure
Time Frame: 12 months post-index procedure
Population: Primary Target Lesion Patency (TLP) at 12 months post-index procedure.
Measure: Number; unit: percentage of participants
Arm/Group | PTA and Study Stent
Number analyzed (Participants) | 65
percentage of participants | 81.5

ADVERSE EVENTS:
Time Frame: Throughout follow-up of study period = 36 months
Arm/Group | PTA and Study Stent
All-Cause Mortality (participants affected / at risk) | 8/76
Serious Adverse Events (participants affected / at risk) | 49/76
Other Adverse Events (participants affected / at risk) | 70/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTA and Study Stent (N=76)
Other (Cardiac disorders) | 14 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Acute Myocardial Infarction (Cardiac disorders) | 2
Angina Pectoris (Cardiac disorders) | 2
Arterial Fibrillation (Cardiac disorders) | 2
Cardiac Failure (Cardiac disorders) | 3
Myocardial Infarction (Cardiac disorders) | 2
Other (Gastrointestinal disorders) | 5 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Inguinal Hernia (Gastrointestinal disorders) | 2
Other (Injury, poisoning and procedural complications) | 19 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Arterial Restenosis (Injury, poisoning and procedural complications) | 2
In-stent Arterial Restenosis (Injury, poisoning and procedural complications) | 16
Other (Musculoskeletal and connective tissue disorders) | 3 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Other (Respiratory, thoracic and mediastinal disorders) | 5 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Dyspnea (Musculoskeletal and connective tissue disorders) | 2
Other (Vascular disorders) | 22 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Arterial restenosis (Vascular disorders) | 3
Arterial restenosis limb (Vascular disorders) | 2
Femoral arterial stenosis (Vascular disorders) | 6
Femoral Arterial Occlusion (Vascular disorders) | 5
Iliac Artery Stenosis (Vascular disorders) | 4
In-stent arterial restenosis (Vascular disorders) | 3
Peripheral arterial occlusive disease (Vascular disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTA and Study Stent (N=76)
Other (Vascular disorders) | 40 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Arterial restenosis (Vascular disorders) | 4
Arterial stenosis lim (Vascular disorders) | 3
Femoral arterial stenosis (Vascular disorders) | 14
Femoral artery occlusion (Vascular disorders) | 6
Hematoma (Vascular disorders) | 4
Iliac artery stenosis (Vascular disorders) | 5
Intermittent claudication (Vascular disorders) | 8
Peripheral arterial occlusive disease (Vascular disorders) | 9
Other (Respiratory, thoracic and mediastinal disorders) | 10 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Other (Musculoskeletal and connective tissue disorders) | 24 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Other (Injury, poisoning and procedural complications) | 35 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Arterial restenosis (Injury, poisoning and procedural complications) | 4
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 18
Post -procedural hematoma (Injury, poisoning and procedural complications) | 15
Other (Infections and infestations) | 9 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Pneumonia (Infections and infestations) | 3
Other (General disorders) | 11 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Pyrexia (General disorders) | 3
Other (Cardiac disorders) | 15 — This includes all AEs in the system organ class (SOC) that were reported by less than two subjects.
Angina pectoris (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No